CLINICAL TRIAL: NCT04875247
Title: IOLMASTER 700 Central Topography Workflow Study.
Status: Completed | Type: Observational
Sponsor: OFTALVIST (Oftalmología Vistahermosa S.L) (Industry)
Responsible Party: Sponsor
Other Study IDs: IOLWORK
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: All patients will be assigned to this cohort.
  Interventions: Device: IOLMaster 700 with central topography; Device: IOLMaster 700 without central topography plus Cassini; Device: IOLMaster 700 without central topography plus Pentacam

INTERVENTIONS:
Device: IOLMaster 700 with central topography — The time needed to perform the measurement using the IOLMaster700 equipment with central topography will be recorded.
Device: IOLMaster 700 without central topography plus Cassini — The time needed to perform the measurement using the IOLMaster700 equipment without central topography plus the Cassini equipment will be recorded.
Device: IOLMaster 700 without central topography plus Pentacam — The time needed to perform the measurement using the IOLMaster700 equipment without central topography plus the Pentacam equipment will be recorded.

SUMMARY:
The use of ocular biometers like IOLMaster 700, is a common practice to identify several ocular parameters such as the keratometry of the cornea and the axial length of the eye, which are necessary for calculating the power of the intraocular lens in cataract surgery. However, the additional use of other devices, such as Cassini and Pentacam is used to obtain more information of the central topography of the eye. Recently, a new version of the IOLMaster 700 equipment that provides much more detailed information than in its previous version has been presented. The objective of this study is to measure the time that the new IOLMaster 700 takes to perform these measurements of the central topography and compare it with the time it takes using the central topography using the standard IOLMaster 700 version with Cassini on one hand and Pentacam on the other.

It is hypothesized that the use of the new version of the IOLMaster 700 equipment alone can reduce the time of measurements and improve the clinic workflow.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have to undergo a cataract surgery
* Patients older than 50 years.

Exclusion Criteria:

* Patients that have already undergone a previous corneal surgery.
* Patients suffering from keratoconus.
* Patients exhibiting corneal scars
* Patients exhibiting pterygium

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 50 years with cataracts that have to undergo a cataracts surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Time needed to do the measurements with each equipment | 1 day (Cataract pre-surgery visit)
  Time needed to do the measurements with each equipment

SECONDARY OUTCOMES:
Central topography | 1 day (Cataract pre-surgery visit)
  Measurement of keratometry (K): Flat Keratometry (K1) and Steep Keratometry (K2)

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Ruiz Mesa., Doctor, Principal Investigator — OFTALVIST (Oftalmología Vistahermosa S.L)
Locations (1):
- OFTALVIST (Oftalmología Vistahermosa S.L.), Jeréz de La Frontera, Cádiz, Spain

REFERENCES:
- [Result] Ruiz-Mesa R, Ruiz-Santos M, Blanch-Ruiz J, Jimenez-Nieto A. Acquisition Time for Swept-Source Optical Biometry Plus Corneal Power Measurement During Cataract Evaluation. Clin Ophthalmol. 2022 Mar 5;16:661-668. doi: 10.2147/OPTH.S351845. eCollection 2022. PMID 35282169